CLINICAL TRIAL: NCT02450682
Title: Evaluate the Safety of Apixaban in Patients Who Undergo Cardiovascular Implantable Electronic Device (CIED) Procedure: A Randomized Pilot Study
Brief Title: Apixaban in Patients Who Undergo CIED Procedure- Randomized Pilot Study
Acronym: Apixaban
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Yong-Mei Cha, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 14-005395
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — apixaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apixaban (Active Comparator): 30 participants prescribed Apixaban 3-14 days before and 28 days after CIED procedure.
  Interventions: Drug: Apixaban
- Warfarin (Other): 30 participants will take stable dose of warfarin and go through the procedure without drug interrupt. The dose is adjusted by INR level. Length of treatment is 42 days, 14 days before and 28 days after the procedure.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Apixaban — Anticoagulant agent for Atrial Fibrillation and undergo CIED generator change
  Other Names: Eliquis
  Arms: Apixaban
Drug: Warfarin — Anticoagulant agent for Atrial Fibrillation and undergo CIED generator change
  Other Names: Coumadin
  Arms: Warfarin

SUMMARY:
This study is being done to determine if apixaban is more safe, when compared to warfarin, at reducing the risk of bleeding during CIED procedures.

ELIGIBILITY:
1. Signed informed written consent
2. Patients are taking warfarin or apixaban chronically
3. Patients are at risk of stroke or systemic embolism
4. Patients have NVAF
5. Patients will undergo CIED generator change
6. Age 18-90
7. Either gender
8. All eligibility criteria must be met

Exclusion:

1. Patient is critically ill, or in unstable condition
2. Patient is at high risk for bleeding, HAS-BLED score ≥ 3
3. Patient is required to take dual antiplatelet agents in addition to anticoagulant drug. (e.g. recent cardiac stent placement)
4. Patients have mechanical cardiac valve or another condition other than NVAF that requires chronic anticoagulation
5. Women of childbearing potential with positive pregnant test
6. Bilirubin >2x upper limit of normal, in association with AST/ALT/ALP >3x upper limit normal
7. Allergy to apixaban and warfarin
8. Subjects requiring taking strong dual inhibitors of CYP3A4 and P-gp who already meet the criteria to take 2.5 mg apixaban
9. Subjects requiring taking strong dual inducers of CYP3A4 and P-gp (.e.g., rifampin, carbamazepine, phenytoin, St. John's wort)
10. Patients who take any investigational drugs within 30 days of enrolling in study.
11. Prisoners or subjects who are involuntarily incarcerated.
12. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2017-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
decrease in the hemoglobin level of 2 g per deciliter or more | 2 months
  Assess the risk of major bleeding when continuing apixaban through the procedure as compared to Warfarin.

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Mei Cha, MD, Principal Investigator — Mayo Clinic; Samuel Asirvatham, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States